CLINICAL TRIAL: NCT03048786
Title: Mobile-based Peer Mentoring for Smoking Cessation: A Pilot Study
Brief Title: Mobile-based Peer Mentoring for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Cancer Society, Inc. (Other); George Washington University (Other); London School of Economics and Political Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 16-18577
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Smoking Cessation; Tobacco Use
Keywords: Peer mentoring; social support; text messaging; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Tobacco Use

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): Participants will receive automated text messages drawn from the script used by SmokefreeTXT.
  Interventions: Behavioral: Control
- Peer Mentoring Arm (Experimental): Participants will receive a modified version of the automated text messages sent to the control arm plus random assignment to a peer mentor.
  Interventions: Behavioral: Peer Mentoring

INTERVENTIONS:
Behavioral: Control — Participants will receive automated text messages used by SmokefreeTXT. The messages are designed to provide encouragement, support, and information about quitting smoking. Participants will receive 1-5 automated messages per day for 6-8 weeks depending on choice of quit date.
  Arms: Control Arm
Behavioral: Peer Mentoring — Participants will receive a modified version of the automated text messages sent to the control arm plus random assignment to a peer mentor. The modified messages include automated "conversation starters," designed to stimulate conversation with the peer mentor. The peer mentor will then send personalized, tailored responses. The peer mentor is a former smoker who has completed a training program developed by the investigator team. Participants will receive 1-5 automated messages per day for 6-8 weeks depending on choice of quit date.
  Arms: Peer Mentoring Arm

SUMMARY:
Despite the availability of a variety of effective treatments for smoking cessation, uptake of treatments is low. The increasing use of smartphone technology presents an exceptional opportunity to expand access to low-cost smoking cessation services. In this pilot study, the investigators will use a text-messaging platform to test peer mentoring for smoking cessation, delivered by former smokers. While peer mentoring is a common approach to health behavior change, it has rarely been used to maximum effect by smoking cessation programs. The text-messaging platform serves as the basis for a randomized controlled trial to test the effectiveness of peer mentoring for smoking cessation.

This pilot will include approximately 200 U.S. adult smokers who will be randomly assigned to a peer mentor or not. Participants in the control group will receive automated text messages used in SmokefreeTXT, a nationwide text-messaging service sponsored by the National Cancer Institute (NCI) in which users receive one to five automated messages per day for up to eight weeks. Smokers in the intervention group will receive a modified version of the same automated messages from SmokefreeTXT, but with additional personalized messages from an assigned peer mentor. Mentors will provide responses to specific questions or comments a smoker may have after receiving the automated messages.

The intervention will last 8 weeks. The study includes primary outcomes to measure the acceptability, engagement, user experience, and early efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Current resident of the U.S.
* Smoked 100 or more cigarettes in lifetime
* Current cigarette smoker
* Access to a device that can take pictures to be uploaded to a website
* Willing to complete a salivary cotinine test

Exclusion Criteria:

* Not a current user of nicotine replacement therapy
* Not a current user of electronic cigarettes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Saliva test for cotinine | 3 months after quit day
  The primary measure of early efficacy is the 7-day point prevalence of abstinence measured 3 months after the quit day, using a saliva cotinine test. The saliva test results will be recorded through a series of photographs and shared with the study team via email or online upload. Participants who self-report having smoked in the last 7 days, as part of the follow-up survey, will be considered to be continuing smokers.

SECONDARY OUTCOMES:
Self-reported smoking status | 3 months after quit day
  Participants will self-report 7-day point prevalence of abstinence in the follow-up survey, measured 3 months after the quit day.
Duration of engagement | Up to 8 weeks
  The primary measure of participant engagement is the number of days from enrollment since the participant last replied to a message asking about the person's status (e.g., mood and cravings). The status messages are common to the scripts sent to participants in the control and peer mentoring arms.
Satisfaction with the program | 3 months after quit day
  The primary measure of acceptability of the intervention is the self-reported rating of participants to the statement, "I liked participating in the iQuit Project." Responses will be on a 5-point Likert scale from "completely disagree" to "completely agree."
Proportion of participants who correctly self-report their message type | 3 months after quit day
  The primary measure of user experience in the intervention is whether participants correctly identify the type of messages they received: automated or personal from a mentor. The measure has four categories:
  1. assigned to automated messages and self-reports receiving automated messages only,
  2. assigned to automated messages and self-reports receiving at least some messages from a mentor,
  3. assigned to mentor messages and self-reports receiving at least some mentor messages, and
  4. assigned to mentor messages and self-reports receiving automated messages only.
Change in average cigarettes per day | 3 months after quit day
  This measures the difference in self-reported average number of cigarettes smoked per day from the baseline survey to the follow-up survey 3 months after quit day
Number of participant messages sent | Throughout the 6-8 week intervention
  This measure of engagement is the number of resp days from enrollment since the participant last replied to a message asking about the person's status (e.g., mood and cravings). The status messages are common to the scripts sent to participants in the control and peer mentoring arms.
Proportion who unsubscribe | Throughout the 6-8 week intervention
  This measure of engagement is the proportion of participants who unsubscribe from the text-messaging intervention prior to the end of the intervention period.
Accuracy of beliefs about personal content | Throughout the 6-8 week intervention
  This is the difference between the percentage of messages reported to be from a mentor (as opposed to being automated) and the actual percentage.

OTHER OUTCOMES:
Self-reported smoking status during the intervention | From quit day to day 90
  This is self-reported 7-day point prevalence based on text message replies to a status message. The status messages were sent at days 7, 14, 21, 28, 35, 42, 60, and 90, relative to the person's quit date.
Recommends the program | 3 months after quit day
  This is a 5-point Likert scale response to "I would recommend the iQuit Project to a friend," assessed in the follow-up survey.
Helpfulness of information | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages contained helpful information on quitting," assessed in the follow-up survey.
Helpfulness in trying to quit | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages helped me try to quit smoking," assessed in the follow-up survey.
Timeliness of messages | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages arrived at the right time," assessed in the follow-up survey.
Personalized content of messages | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages were created for me personally," assessed in the follow-up survey.
Frequency of messages too low | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages should have been sent more frequently," assessed in the follow-up survey.
Frequency of messages too high | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages should have been sent less frequently," assessed in the follow-up survey.
Tailoring of messages | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages applied to me specifically," assessed in the follow-up survey.
Messages were caring | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages made me feel someone cared if I quit," assessed in the follow-up survey.
Messages gave feeling of worth | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages made me think that it was worthwhile for me to quit," assessed in the follow-up survey.
Messages gave feeling of competence | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages made me feel that I knew the right steps to take to quit," assessed in the follow-up survey.
Messages gave feeling of confidence | 3 months after quit day
  This is a 5-point Likert scale response to "Text messages gave me confidence that I can quit," assessed in the follow-up survey.
Days to unsubscribe | Throughout the 6-8 week intervention
  This is the number of days since enrollment that it took the participant to unsubscribe.
Proportion of replies that provide informational vs. emotional support | Throughout the 6-8 week intervention
  This is the proportion of a participant's replies that are in response to a message coded with information support, as opposed to emotional support.
Percentage of personalized messages | 3 months after enrollment
  This is the percentage of messages that the participant believes came from a mentor, as opposed to the automated script.
Preference for personalized messages | 3 months after enrollment
  This is the percentage of participants who prefer personal messages from mentors, compared to automated messages.
Integration of messages | 3 months after enrollment
  This is a 5-point Likert scale response to "The automated and personal messages worked well together," assessed in the follow-up survey.
Satisfaction with mentor | 3 months after enrollment
  This is a 5-point Likert scale response to "I am satisfied with my mentor," assessed in the follow-up survey.
Knowledge of mentor | 3 months after enrollment
  This is a 5-point Likert scale response to "I think my mentor was knowledgable," assessed in the follow-up survey.

CONTACTS AND LOCATIONS:
Overall Officials: Justin S White, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] White JS, Toussaert S, Thrul J, Bontemps-Jones J, Abroms L, Westmaas JL. Peer Mentoring and Automated Text Messages for Smoking Cessation: A Randomized Pilot Trial. Nicotine Tob Res. 2020 Mar 16;22(3):371-380. doi: 10.1093/ntr/ntz047. PMID 30892616